CLINICAL TRIAL: NCT00938184
Title: An Open Label, Randomized, Three-period Crossover Study to Compare the Pharmacokinetic Profile of Paroxetine After Single Doses of the Controlled-release Paroxetine Tablets at the Dose Levels of 12.5, 25 and 50mg in Healthy Japanese Male Subjects
Brief Title: Single Dose Study of Controlled-Release Paroxetine Tablets in Healthy Japanese Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 112811
Record Dates: First submitted 2009-07-09; First posted 2009-07-13 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Depressive Disorder
Keywords: tolerance; single dose; paroxetine; controlled-release tablet; safety; pharmacokinetics; Japanese healthy male subjects
MeSH Terms: conditions — Depressive Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Treatment sequence A/B/C (Experimental): Eligible subjects will be randomized in sequence A/B/C and will receive A: single tablet of paroxetine 12.5 milligrams, B: single tablet of paroxetine 25 milligrams and C: two tablets of paroxetine 25 milligrams administered orally in the morning. Subjects will be fasting since 10 hours before dosing in each period.
  Interventions: Drug: Paroxetine 12.5 milligrams tablet; Drug: Paroxetine 25 milligrams tablet; Drug: Paroxetine 50 milligrams tablet
- Treatment sequence A/C/B (Experimental): Eligible subjects will be randomized in sequence A/C/B and will receive A: single tablet of paroxetine 12.5 milligrams, C: two tablets of paroxetine 25 milligrams and B: single tablet of paroxetine 25 milligrams administered orally in the morning. Subjects will be fasting since 10 hours before dosing in each period.
  Interventions: Drug: Paroxetine 12.5 milligrams tablet; Drug: Paroxetine 25 milligrams tablet; Drug: Paroxetine 50 milligrams tablet
- Treatment sequence B/A/C (Experimental): Eligible subjects will be randomized in sequence B/A/C and will receive B: single tablet of paroxetine 25 milligrams, A: single tablet of paroxetine 12.5 milligrams and C: two tablets of paroxetine 25 milligrams administered orally in the morning. Subjects will be fasting since 10 hours before dosing in each period.
  Interventions: Drug: Paroxetine 12.5 milligrams tablet; Drug: Paroxetine 25 milligrams tablet; Drug: Paroxetine 50 milligrams tablet
- Treatment sequence B/C/A (Experimental): Eligible subjects will be randomized in sequence B/C/A and will receive B: single tablet of paroxetine 25 milligrams, C: two tablets of paroxetine 25 milligrams and A: single tablet of paroxetine 12.5 milligrams administered orally in the morning. Subjects will be fasting since 10 hours before dosing in each period.
  Interventions: Drug: Paroxetine 12.5 milligrams tablet; Drug: Paroxetine 25 milligrams tablet; Drug: Paroxetine 50 milligrams tablet
- Treatment sequence C/A/B (Experimental): Eligible subjects will be randomized in sequence C/A/B and will receive C: two tablets of paroxetine 25 milligrams, A: single tablet of paroxetine 12.5 milligrams and B: single tablet of paroxetine 25 milligrams administered orally in the morning. Subjects will be fasting since 10 hours before dosing in each period.
  Interventions: Drug: Paroxetine 12.5 milligrams tablet; Drug: Paroxetine 25 milligrams tablet; Drug: Paroxetine 50 milligrams tablet
- Treatment sequence C/B/A (Experimental): Eligible subjects will be randomized in sequence C/B/A and will receive C: two tablets of paroxetine 25 milligrams, B: single tablet of paroxetine 25 milligrams and A: single tablet of paroxetine 12.5 milligrams administered orally in the morning. Subjects will be fasting since 10 hours before dosing in each period.
  Interventions: Drug: Paroxetine 12.5 milligrams tablet; Drug: Paroxetine 25 milligrams tablet; Drug: Paroxetine 50 milligrams tablet

INTERVENTIONS:
Drug: Paroxetine 12.5 milligrams tablet — Single dose of paroxetine 12.5 milligrams controlled release tablet will be administered orally.
Drug: Paroxetine 25 milligrams tablet — Single dose of paroxetine 25 milligrams controlled release tablet will be administered orally.
Drug: Paroxetine 50 milligrams tablet — Single dose of paroxetine 50 milligrams controlled release tablet (as two tablets of 25 milligrams) will be administered orally.

SUMMARY:
The primary purpose of this study is to to assess the pharmacokinetics of paroxetine after single doses of paroxetine CR at the dose levels of 12.5, 25 and 50mg in healthy Japanese male volunteers.

DETAILED DESCRIPTION:
This clinical trial is to characterize the pharmacokinetic profile after single oral doses of the proposed final market tablet formulations of paroxetine CR in Japan (the 12.5mg and 25mg tablets), at the dose levels of 12.5, 25 and 50mg in the healthy male Japanese volunteers. Treatment sequence of the 3 dose levels in each subject is randomized.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Japanese adult males between 20 and 64 years of age inclusive
* BMI 18.50 or higher and < 25.00 kg/m2, and bodyweight 50 kg or higher
* Non-smokers
* AST, ALT, ALP, gamma-GTP and total-bilirubin are below the upper limit of normal range
* QTc(B) interval <450 msec
* Able to attend all visits and complete the study
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form

Exclusion Criteria:

* Any clinically relevant abnormality on the screening physical examination, vital signs, 12-lead ECG and/or clinical laboratory tests
* Medical history that is not considered as eligible for inclusion in this study by the investigator
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of asymptomatic gallstones)
* History of psychiatric disorder or suicide attempts or behaviours
* History or presence of gastrointestinal, hepatic or renal disease or any other condition known to interfere with the absorption, distribution, metabolism or excretion of drugs
* History of sensitivity to any of the paroxetine formulations, or components thereof
* Positive for urine drug screening
* Participation in another clinical study or post-marketing study in which the subject is or will be exposed to an investigational or a non-investigational product or device
* Participation in a clinical study or post-marketing study with an investigational or a non-investigational product or device within 4 months of preceding the first dose of study medication
* History of drug or other allergy, or idiosyncrasy, excluding a pollen allergy without current symptoms
* History of drug abuse, or current conditions of drug abuse or alcoholism
* History of regular alcohol consumption exceeding, on average, 14 drinks/week (1 drink = 150 mL of wine or 350 mL of beer or 45 mL of 80 proof distilled spirits) within 6 months of screening
* Use of prescription or no-prescription drugs, including vitamins, crude drug, herbal and dietary supplements (including St John's Wort) within 14 days prior to the first dose of study medication
* Unwillingness or inability to follow the procedures outlined in the protocol
* Consumption of grapefruit or grapefruit-containing products from 7 days prior to the first dose of study medication
* Positive for syphilis, HIV antibody and antigen, Hepatitis B surface antigen, Hepatitis C antibody or HTLV-1 antibody
* Donation of blood in excess of 400mL within the previous 4 months or 200mL within the previous 1 month to the first dose of study medication

Ages: 20 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2009-07-14 (Actual); Primary Completion 2009-09-02 (Actual); Study Completion 2009-09-02 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters of plasma paroxetine after single doses of paroxetine CR at 12.5mg, 25mg and 50mg in healthy Japanese male volunteers | up to 120 hours after a single dose in all dosing sessions

SECONDARY OUTCOMES:
Safety and tolerability after single doses of paroxetine CR at 12.5mg, 25mg and 50mg in healthy Japanese male volunteers | up to 120 hours after a single dose in all dosing sessions

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study 112811 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/112811?search=study&study_ids=112811#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 112811 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 112811 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 112811 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 112811 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register